CLINICAL TRIAL: NCT00386789
Title: Long Term Protection by and Persistence of Vi Antibodies Induced by Vi-rEPA Conjugate Vaccines in Vietnamese Children Injected at 2-5 Years or at 5-8 Years of Age
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907004; 07-CH-N004
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Typhoid Fever
Keywords: Typhoid Fever; Serological Survey; Follow-Up; Protection
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Typhoid fever remains an important cause of morbidity and mortality in the developing world. It is estimated that more than 16 million cases and about 600,000 deaths occur annually, most of which occur in Southeast Asia and Africa. Ingestion of food or water contaminated by acutely infected persons or chronic carriers is the most common form of transmission. As a result, typhoid fever is prevalent where unsafe drinking water or contaminated food is common.

Typhoid fever is highly endemic in Vietnam, especially in the southern provinces and is a significant disease in both preschool and school-aged children. Data from Dong Thap Provincial Hospital, Mekong delta region showed that among 3,934 hospitalized typhoid fever cases from 1990 to 1995, 4.2% had complications and 0.8% died.

Typhoid fever has become difficult and expensive to treat. About 90% of Salmonella typhi isolates are of multidrug-resistant (resistant to chloramphenicol, ampicillin, and trimethoprim-sulfamethoxazole) and 76% of isolates showed reduced susceptibility to fluoroquinolones. Isolates with full fluoroquinolone or extended spectrum cephalosporin resistance have not yet reported in Vietnam but occur sporadically in the Indian subcontinent. If they become widespread, alternative treatment options will be limited. The improvement of sanitation, provision of safe water and elimination of chronic carriage is not expected to be achieved quickly. Accordingly, vaccination against typhoid fever is increasingly important national public health priority.

DETAILED DESCRIPTION:
Typhoid fever remains an important cause of morbidity and mortality in the developing world. It is estimated that more than 16 million cases and about 600,000 deaths occur annually, most of which occur in Southeast Asia and Africa. Ingestion of food or water contaminated by acutely infected persons or chronic carriers is the most common form of transmission. As a result, typhoid fever is prevalent where unsafe drinking water or contaminated food is common.

Typhoid fever is highly endemic in Vietnam, especially in the southern provinces, and is a significant disease in both preschool and school-aged children. Data from Dong Thap Provincial Hospital, Mekong delta region showed that among 3,934 hospitalized typhoid fever cases from 1990 to 1995, 4.2% had complications and 0.8% died.

Typhoid fever has become difficult and expensive to treat. About 90% of Salmonella typhi isolates are of multidrug-resistance (resistant to chloramphenicol, ampicillin, and trimethoprim-sulfamethoxazole) and 76% of isolates showed reduced susceptibility to fluoroquinolones. Isolates with full fluoroquinolone or extended spectrum cephalosporin resistance have not been reported yet in Vietnam but occur sporadically in the Indian subcontinent. If they become widespread, alternative treatment options will be limited. The improvement of sanitation, provision of safe water and elimination of chronic carriage are not expected to be achieved quickly. Accordingly, vaccination against typhoid fever is an increasingly important national public health priority.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who were involved in the Phase III trial, OH98-CH-N002.

EXCLUSION CRITERIA:

Not specified.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0
Dates: Start 2006-10-05; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (4):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States
- Vietnam (3):
  - Dong Thap Provincial Hospital, Dong Thập
  - National Institute of Hygiene and Epidemiology, Hanoi
  - Pasteur Institute, Ho Chi Minh City

REFERENCES:
- [Background] Smith MD, Duong NM, Hoa NT, Wain J, Ha HD, Diep TS, Day NP, Hien TT, White NJ. Comparison of ofloxacin and ceftriaxone for short-course treatment of enteric fever. Antimicrob Agents Chemother. 1994 Aug;38(8):1716-20. doi: 10.1128/AAC.38.8.1716. PMID 7986000